CLINICAL TRIAL: NCT07087392
Title: Modified Digestive Tract Reconstruction in Laparoscopic Duodenum-Preserving Pancreatic Head Resection or Laparoscopic Central Pancreatectomy: Inverted-Ω Anastomosis
Brief Title: Inverted-Ω Anastomosis in Laparoscopic Duodenum-Preserving Pancreatic Head Resection or Laparoscopic Central Pancreatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-550
Record Dates: First submitted 2025-07-08; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cystic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inverted-Ω Anastomosis (Experimental): After meeting the inclusion and exclusion criteria, duodenum-preserving pancreatic head resection or mid-pancreatic resection will be performed, and inverted-Ω anastomosis will be carried out during the operation for the reconstruction of the digestive tract
  Interventions: Procedure: Inverted-Ω Anastomosis

INTERVENTIONS:
Procedure: Inverted-Ω Anastomosis — After meeting the inclusion and exclusion criteria, duodenum-preserving pancreatic head resection or mid-pancreatic resection will be performed, and inverted-Ω anastomosis will be carried out during the operation for the reconstruction of the digestive tract

SUMMARY:
The goal of this clinical trial is to learn if inverted-Ω anastomosis after pancreatic head resection or mid-pancreatectomy works in benign or low-grade malignant tumor. It will also learn about the safety and feasibility of inverted-Ω anastomosis. The main questions it aims to answer are:

1. Does inverted-Ω anastomosis operate safely? (operative time, blood loss, transfusion and conversion rate)
2. What is the incidence and severity of postoperative complications in inverted -Ω anastomosis? What advantages does it have over conventional anastomosis methods such as roux-en-y？

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old, gender not limited;
2. Patients diagnosed with benign or low-grade malignant tumors in the head or middle section of the pancreas by CT or MRI;
3. ECOG score 0-1.

Exclusion Criteria:

1. Those with severe heart, liver or kidney insufficiency, or those who are assessed as intolerant to surgery or anesthesia, or those with ASA grade > 3;
2. Patients with a history of or concurrent other malignant tumors, or other serious infections or infectious diseases, or those who are unable to complete the anastomosis surgery;
3. Uncontrollable concomitant diseases, including but not limited to severe coronary artery disease, COPD or asthma, uncontrollable cerebrovascular diseases, symptomatic congestive failure, unstable angina pectoris, arrhythmia, or other diseases that the researchers consider ineligible for enrollment;
4. Patients who have undergone other upper abdominal surgeries and digestive tract reconstruction procedures in the past;
5. Patients requiring combined organ resection;
6. Preoperative assessment suggested that the patient might have factors such as active ulcers and bleeding in the digestive tract;
7. Pregnant and lactating women;
8. Any uncertain factors that have an impact on the patient's safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2028-07-20 (Estimated)

PRIMARY OUTCOMES:
Safety and assessment of the surgical process | During operation
  The incidence of intraoperative adverse events such as conversion to open surgery rate
Operative time | During operation
  Operative time
Intraoperative blood loss | During operation
  Intraoperative blood loss
Postoperative complications | From the date of surgery (Day 0) up to 90 days postoperatively
  The incidence and severity of postoperative complications, as defined by the International Study Group on Pancreatic Surgery (ISGPS)

SECONDARY OUTCOMES:
Short-term survival | From the date of surgery (Day 0) up to 3 years postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No